CLINICAL TRIAL: NCT02429128
Title: 14 Weeks Exercise Training on Lean Women With and Without PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Solvejg Hansen, Cand Scient Human Physiology, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Lean PCOS & Training
Record Dates: First submitted 2015-04-15; First posted 2015-04-29 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean PCOS training (Active Comparator): 14 weeks exercise training
  Interventions: Other: 14 weeks exercise training
- Lean healthy controls (Other): 14 weeks exercise training
  Interventions: Other: 14 weeks exercise training

INTERVENTIONS:
Other: 14 weeks exercise training

SUMMARY:
The aim of this project is to investigate the pathophysiology of PCOS in regards to the metabolic profile including defects in insulin sensitivity in skeletal muscle and adipose tissue, and to investigate the effects of exercise training on these parameters.

ELIGIBILITY:
Inclusion Criteria: Women with PCOS

* Hyperandrogenism and/or hyperandrogenemia
* Regular menstruation
* Age: 20-40
* Inactive or low physical activity level
* Low to moderate fitness status

Inclusion Criteria: Women without PCOS

* Normal levels of plasma androgens
* Polycystic ovary and/or menstrual dysfunction
* Age: 20-40
* Inactive or low physical activity level
* Low to moderate fitness status

Exclusion Criteria: Women with and without PCOS

* Pregnancy or breast feeding
* Smoking
* Use of birth control pills 3 mo before enrolment

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Compliance to exercise training program as assessed by number of training sessions completed | 14 weeks
  Superviced training program - no. of training sessions are noted by trainer. Compliance must be higher than 80%.
No change in Body Weight | 14 weeks
Component of metabolic syndrome | 14 weeks
  Hole body insulin sensitivity measured by HOMA index
Component of metabolic syndrome | 14 weeks
  Peripheral insulin sensitivity measured by hyperinsulinemic euglycemic clamp methods.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, Professor, Study Director — NEXS, KU
Locations (1):
- August Krogh Building, Copenhagen, Østerbro, Denmark

REFERENCES:
- [Derived] Hansen SL, Svendsen PF, Jeppesen JF, Hoeg LD, Andersen NR, Kristensen JM, Nilas L, Lundsgaard AM, Wojtaszewski JFP, Madsbad S, Kiens B. Molecular Mechanisms in Skeletal Muscle Underlying Insulin Resistance in Women Who Are Lean With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2019 May 1;104(5):1841-1854. doi: 10.1210/jc.2018-01771. PMID 30544235